CLINICAL TRIAL: NCT06237140
Title: Comparison of the Effectiveness of Cervical Proprioceptive Neuromuscular Facilitation and Stabilization Exercises on Balance, Fall Risk and Fear of Falling in Stroke Patients
Brief Title: Cervical Proprioceptive Neuromuscular Facilitation and Stabilization Exercises in Stroke Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was registered in error.
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Güler ERTUĞRUL, MSc student, physiotherapist, Suleyman Demirel University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 791
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Stroke
Keywords: proprioception; stabilization exercises; balance; fall
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomization order tracking will be done with sequentially numbered containers. Patients participating in the study will be blinded to which treatment group they will be included in.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients participating in the study will be blinded to which treatment group they will be included in. The evaluations of the patients participating in the study will be evaluated by a physiotherapist who is blind to group assignments. During treatment, physical therapists will be instructed not to communicate with patients about the possible goals or rationale for either treatment. A professional who is blind to the evaluation results of the groups will perform the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF exercise group (Experimental): proprioceptive neuromuscular facilitation (PNF) techniques will be applied to the cervical region. In the study, flexion-lateral flexion and rotation patterns will be studied together with antagonist patterns. In the antagonist movement involving cervical extension, the hand above the head is displaced diagonally and positioned to resist extension, lateral flexion and rotation. Before the exercise, the patient will be informed about the diagonal direction of the movement and made to feel it, and then the exercises will be performed in 5 sets, each set containing 10 repetitions. Participants will be given sufficient time to rest between sets.
  Interventions: Other: PNF+ biofeedback exercise group
- biofeedback exercise group (Active Comparator): cervical stabilization exercises will be used to stimulate cervical proprioceptors. Neck stabilization training will be applied with a low load to strengthen the longus capitis and longus colli, the deep muscles of the upper cervical vertebra. The oblique and costal muscles, which are the auxiliary respiratory muscles, will be relaxed and the neck will be flexed. A pressure biofeedback device will be placed on the upper cervical spine (below the occiput) while lying with the air pocket set at 20 mmHg to obtain visual feedback from the dial. The pressure will be gradually increased to 30 mmHg in 2 mmHg increments. While the patient was asked to retract his chin, the contraction duration was determined as 10 seconds. While the contractions are repeated 10 times, a 3-5 second rest period will be given between each contraction.
  Interventions: Other: PNF+ biofeedback exercise group

INTERVENTIONS:
Other: PNF+ biofeedback exercise group — Neurorehabilitation will be applied to this group, 5 sessions a week for 4 weeks, to increase balance and walking skills and reduce the risk of falling.

SUMMARY:
Randomization order tracking will be done with sequentially numbered containers. Patients participating in the study will be blinded as to which treatment group they will be included in. Before the study, written and verbal "Informed Consent Form" will be obtained from all participants who meet the inclusion criteria. In order to prevent bias, participants assigned to groups will be evaluated by a blind physiotherapist. Tests; The treatment of patients in the study and control groups will be carried out one day before the start, and all evaluations will be repeated after the 4-week neurorehabilitation process is completed. All data obtained will be noted on the prepared evaluation form.

DETAILED DESCRIPTION:
Randomization order tracking will be done with sequentially numbered containers. Patients participating in the study will be blinded to which treatment group they will be included in. Before the study, written and verbal "Informed Consent Form" will be obtained from all participants who meet the inclusion criteria. After the sociodemographic and clinical features of the participants are recorded, the cognitive status of the patients will be evaluated with MMT. Participants' neck proprioceptive senses, cervical proprioceptive awareness, cervical joint failure test, falling risks, dynamic and static balance tests on the Tecnobody Prokin 252 Isokinetic Balance Platform, among objective tests, Timed up and go test and Berg balance test, among clinical tests, and their fear of falling, Modified. It will be evaluated with the Fall Effectiveness Scale. To avoid bias, evaluations will be made by a blind physiotherapist to the participants assigned to the groups. Tests; It will be done one day before the treatments to the patients in the study and control groups begin, and all evaluations will be repeated after the 4-week neurorehabilitation process is completed. All data obtained will be noted on a prepared evaluation form.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Volunteering to participate in the study
* Being between the ages of 35-75
* Being diagnosed with stroke
* Having a stroke for the first time
* Mini Mental Test (MMT) Score ≥ 24
* Brunnstorm lower extremity stage ≥ 2
* Being clinically stable

Exclusion Criteria:

* Mini Mental Score < 24 points
* Having additional hearing and vestibular system problems
* Having problems with field of vision
* Orthopedically sourced platinum etc. on his body. having had an operation
* Having a cerebrum, cerebellar or spinal cord malignancy
* Having additional neurological lesions (MS, Parkinson's, Alzheimer's)
* Mini Mental Score < 24 points
* Having cervical pain of 5 or higher on the visual analog scale
* Having serious vestibular, auditory and visual problems that affect balance (vertigo, etc.)
* Having a history of orthopedic surgery for the trunk and lower extremities
* Presence of an additional neurological disease (MS, Parkinson's, Alzheimer's)
* Having joint rigidity that prevents proprioceptive evaluation

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Mini Mental Test | four weeks
  It will be used to evaluate the cognitive status of patients. It is a simple, short and valid test that is widely used in stroke patients. With this test, various cognitive functions of people such as orientation, recording memory, attention and calculation, recall and language are evaluated. The maximum score that can be obtained from the test is 30. Getting a score of 24 or above indicates that the patient's cognitive functions are within normal limits.
cervical joint position error test | four weeks
  In this test, the laser pointer on the helmet and the circle shown at 1 cm intervals are used as a target board. Patients are seated in a chair with back support, 90 cm away from the target board fixed to the wall. Patients are first asked to memorize the position of their head without leaning in any direction and try to find the same point after an active head movement. Active head movements include flexion, extension, and right and left rotations. The desired movements are repeated 10 times. After the movement, the horizontal, vertical and global distances of each point returned to the starting point will be recorded. To calculate the test result, the average values of the incorrect distances in centimeters will be calculated.
Tecnobody Prokin 252 balance platform | four weeks
  To measure balance performance, patients are given the Tecnobody Prokin 252 balance platform. The moving balance platform works with air piston servo motors. Thanks to the automatic engine locking function, the system instantly switches from dynamic measurement to static measurement and provides measurement of two different balances with objective results.
Berg Balance Scale | four weeks
  Berg Balance Scale (BDI) is a scale that contains 14 instructions and scores between 0-4 are given by observing the patient's performance for each instruction. A score of 0 is given when the patient cannot do the activity at all, while a score of 4 is given when the patient completes the activity independently. The highest score is 56, 0-20 points indicate imbalance, 21-40 points indicate acceptable balance, and 41-56 points indicate good balance. It takes between 10 and 20 minutes to complete the scale.
Timed-Up and Go Test | four weeks
  It is one of the most frequently preferred evaluation methods as it is a test that includes movement maneuvers used in daily life. The test begins with a sitting position on a chair. The person is asked to get up from the chair he/she is sitting on, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair again. The time it takes to complete the test is recorded in seconds. While healthy individuals generally complete the test in less than 10 s, individuals who complete it in more than 30 s are classified as dependent on many activities of daily life and mobility skills.
Modified Fall Activity Scale | four weeks
  14 items (10 indoor and 4 outdoor activities) assess confidence when performing different daily tasks. Items on the scale are scored from 0 (unsafe) to 10 (completely safe) to rate participants' level of fall-related self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLER ERTUĞRUL, Principal Investigator — Süleyman Demirel University Faculty of Health Sciences
Locations (1):
- Güler Ertuğrul, Kocaeli, Gölcük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No